CLINICAL TRIAL: NCT01328977
Title: Trial to Assess Best Methods for Engaging Academic Physicians in Grateful Patient Philanthropy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NA_00029824
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Physician's Role
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- emails, book (Active Comparator)
  Interventions: Behavioral: education
- didactic teaching from experts (Active Comparator)
  Interventions: Behavioral: education
- personal coaching by development profs (Experimental)
  Interventions: Behavioral: education

INTERVENTIONS:
Behavioral: education — teaching

SUMMARY:
This study attempted to identify the best method for educating and engaging academic physicians in grateful patient philanthropy.

DETAILED DESCRIPTION:
In this small trial assessing the impact of educational methodologies, we are looking to determine which of the following 3 approaches will be most successful in engaging academic physicians in grateful patient philanthropy;

* email advice
* didactic session led by experts
* one-on-one coaching by development professionals

ELIGIBILITY:
Inclusion Criteria:

* academic physicians

Exclusion Criteria:

* having secured grateful patient philanthropy in past

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
qualified referrals to development office | 6 month follow-up period
  Individuals able to make a donation of $25,000 based on criteria established by Hopkins Office of Development.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Wright, MD, Principal Investigator — JHU SOM